CLINICAL TRIAL: NCT06705387
Title: DeTECTS: Dupilumab Versus Topical Corticosteroid Effectiveness - Comparison in the Treatment of Stenotic EoE
Brief Title: Dupilumab Versus Topical Corticosteroid Effectiveness - Comparison in the Treatment of Stenotic EoE
Acronym: DeTECTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-2367; 1R01DK135692-01A1 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-11-26 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: Dupilumab; Fluticasone
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dupilumab (also known as Dupixent) (Active Comparator)
  Interventions: Biological: Dupilumab
- fluticasone (also known as Flovent) (Active Comparator)
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Biological: Dupilumab — Subcutaneous injection of 300mg per week for 16 weeks.
  Other Names: Dupixent
  Arms: dupilumab (also known as Dupixent)
Drug: Fluticasone — Metered dose swallowed topical corticosteroid, given 1760mcg per day for 16 weeks.
  Other Names: Flovent
  Arms: fluticasone (also known as Flovent)

SUMMARY:
The goal of this clinical trial is to [primary purpose: e.g., learn if intervention or health behavior can treat, prevent, diagnose etc.] in [describe participant population/primary condition; could include any of the following: sex/gender, age groups, healthy volunteers]. The main question[s] it aims to answer [is/are]:

Does dupilumab or swallowed topical fluticasone improve the diameter of the esophagus more? Does dupilumab or swallowed topical fluticasone reduce inflammation in the esophagus more? Are comparative effective clinical trials feasible in this patient population?

Researchers will compare dupilumab 300 mg weekly compared to swallowed fluticasone to see if there is a difference in treatment response.

Participants will be asked to:

* Be randomized to either dupilumab sq weekly or swallowed topical fluticasone twice daily.
* Participate in 8 study visits over 52 weeks
* Complete questionnaires
* Have an endoscopy with biopsies and EndoFLIP measurements.
* Swallow an Esophageal String Test

ELIGIBILITY:
Inclusion Criteria:

* Seen at CHCO for clinical care.
* Age 12 - 25 years old inclusive
* Weight ≥40 kg at the time of screening visit
* Confirmed EoE as diagnosed by biopsy with eosinophils ≥15 eosinophils/hpf in at least 2 esophageal regions at screening endoscopy
* Report of an average of at least 2 episodes of dysphagia per week in the 4 weeks prior to screening.
* Evidence of fibrostenotic features at time of screening endoscopy (grade 2 or 3 esophageal rings, stricture, delayed passage of barium tablet on fluoroscopy, and/or distensibility ≤15mm)

Exclusion Criteria:

* Esophageal dilation performed at index endoscopy
* Patients with stricture undergoing dilation at index endoscopy may be rescreened if they meet all other eligibility criteria.
* Patients with acute food impaction will not be enrolled at their therapeutic endoscopy but are eligible for enrollment subsequently if they meet all other eligibility criteria.
* Eligible patients on current STCs can be enrolled but need to be on stable dosing less than or equal to 440 mcg two times daily fluticasone equivalent for 3 months prior to enrollment.
* Patients who have received dupilumab in the past 12 months for any indication are excluded.
* Diet restrictions and PPI use must stay unchanged in the 8 weeks prior to index endoscopy and through the study period.
* Patients with a fasting morning cortisol <5 within 2 months of screening will not be enrolled. If repeat cortisol levels are normal, patients can be reconsented.
* Known other esophageal disease or esophageal injury (e.g. achalasia, tracheoesophageal fistula, congenital stricture, caustic injury, history of esophageal surgery), inflammatory bowel disease, liver disease, connective tissue disorder, or bleeding disorder.
* Patients with a known gelatin allergy will be excluded from EST collection.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Esophageal Lumen Distensibility | From baseline endoscopy to the end of treatment at week 16.
  Change in distensibility (mm) from baseline to end of treatment (continuous). This is measured by EndoFLIP.
Reduction of epithelial eosinophilia to < 15 eos/hpf (binary) | This will be measured at week 16 end of treatment.
  The number of patients meeting a reduction in epithelial eosinophilia on esophageal biopsies of <15 eos/hpf at end of treatment.

SECONDARY OUTCOMES:
Change in daily symptom questionnaire (DSQ) severity score | From screening to the end of treatment at week 16.
  The change in daily symptoms as measured by the DSQ severity score from enrollment to end of treatment at week 16. A possible DSQ score can range between 0 and 84.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado/University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No